CLINICAL TRIAL: NCT02092207
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, 12 Weeks, Phase II Clinical Study to Evaluate the Safety and Efficacy of Orally Administered KL7016 in Patients With Dry Eye Syndrome
Brief Title: Phase 2 Study to Evaluation the Safety and Efficacy of Orally Administered KL7016 in Patients With Dry Eye Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KL7016_201
Record Dates: First submitted 2014-03-17; First posted 2014-03-20 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- KL7016 900mg (Experimental)
  Interventions: Drug: KL7016 900mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- KL7016 600mg (Experimental)
  Interventions: Drug: KL7016 600mg

INTERVENTIONS:
Drug: KL7016 900mg — oral administration, 150mg 3tab, bid
  Arms: KL7016 900mg
Drug: KL7016 600mg — oral administration, 150mg 3tab, bid
  Arms: KL7016 600mg
Drug: Placebo — oral administration, 150mg 3tab, bid
  Arms: Placebo

SUMMARY:
This is a controlled study to determine the effectiveness and safety of KL7016 in the treatment of adult patients with dry eye syndrome (DES).

ELIGIBILITY:
Inclusion Criteria:

* Corneal staining score of ≥5 in either eye by the National Eye Institute/Industry Workshop guidelines
* Schirmer test score (without anesthesia) < 7 mm/5 min in either eye
* Willing to use no topical ocular treatments, other than REFRESH TEARS® for the duration of the trial

Exclusion Criteria:

* Intraocular surgery within 3months
* Persistent intraocular inflammation or infection
* Corneal transplantation or neurotrophic keratitis
* Stevens-Johnson Syndrome
* Ocular herpes simplex virus infection
* Concomitant use of contact lenses or use within 3months
* Silicone lacrimal punctal occlusion or cauterization of the punctum within 3months
* Vision correction surgery without DES within 12months
* Unstable use of methotrexate or Disease-modifying drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in corneal staining score | baseline, 12 weeks

SECONDARY OUTCOMES:
Change in schirmer test score | baseline, 4weeks, 8weeks, 12 weeks
Change in OSDI(Ocular Surface Disease Index) | baseline, 4weeks, 8weeks, 12 weeks
Change in TFBUT(Tear Film Break-up Time) | baseline, 4weeks, 8weeks, 12 weeks
Change in conjunctival staining score | baseline, 4weeks, 8weeks, 12 weeks
Change in corneal staining score | baseline, 4weeks, 8weeks

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Banpo-daero, Seocho-gu
  - Gangnam Severance Hospital, Seoul, Eonju-ro, Gangnam-gu
  - Seoul National University Bundang Hospital, Gyeonggi-do, Gumi-ro 173 Beon-gil Bundang-gu
  - Korea University Guro Hospital, Seoul, Gurodong-ro, Guro-gu
  - Samsung Medical Center, Seoul, Irwon-ro, Gangnam-gu
  - Chonnam National University Hospital, Gwangju, Jebong-ro, Dong-gu
  - Konkuk University Medical Center, Seoul, Neungdong-ro, Gwangjin-gu
  - ASAN Medical Center, Seoul, Olympic-ro 43-gil, Songpa-gu
  - Severance Hospital, Seoul, Yonsei-ro, Seodaemun-gu